CLINICAL TRIAL: NCT03073213
Title: A Phase 1, Single- and Multiple-Dose Study to Assess the Safety and Pharmacokinetics of Ixekizumab (LY2439821) (Anti-IL-17 Humanized Antibody) in Chinese Patients With Psoriasis Vulgaris
Brief Title: A Study of Ixekizumab in Chinese Participants With Psoriasis Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15371; I1F-MC-RHBN (Other: Eli Lilly and Company)
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2019-06-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Ixekizumab single dose (Experimental): Participants received single dose of 80mg Ixekizumab by subcutaneous injection.
  Interventions: Drug: Ixekizumab
- Ixekizumab Multiple Regimen 1 (80mg Q2W) (Experimental): Participants received multiple doses of Ixekizumab starting with 160mg initial dose followed by 80mg every two weeks (Q2W) by subcutaneous injection.
  Interventions: Drug: Ixekizumab
- Ixekizumab Multiple Regimen 2 (80mg Q4W) (Experimental): Participants received multiple doses of 80mg Ixekizumab starting with 160mg initial dose followed by 80mg every four weeks (Q4W) by subcutaneous injection.
  Interventions: Drug: Ixekizumab

INTERVENTIONS:
Drug: Ixekizumab — Administered as subcutaneous (SC) injection
  Other Names: LY2439821

SUMMARY:
The purpose of the study is to research how much ixekizumab enters the bloodstream and how long the body takes to get rid of the drug and the safety of ixekizumab and any side effects that might be associated with it. The study has two parts: A single-dose part and multiple-dose part. The single dose part of this study will last up to 24 weeks, including the screening period. The multiple dose part of this study will last up to 32 weeks including the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 years.
* Diagnosis of chronic plaque psoriasis for ≥6 months before baseline.
* Candidates for phototherapy and/or systemic therapy.
* ≥10% body surface area (BSA) involvement at screening and baseline.
* static Physician's Global Assessment (sPGA) score ≥3, and Psoriasis Area and Severity Index (PASI) score ≥12 at screening and baseline.

Exclusion Criteria:

* Clinically significant flare of psoriasis during the 12 weeks before baseline.
* Systemic nonbiologic psoriasis therapy or phototherapy within 4 weeks. prior to baseline or topical psoriasis treatment or medicated shampoo within 2 weeks prior to baseline .
* Current or recent use of any biologic agent within the required washout periods.
* Clinical evidence or suspicion of active tuberculosis or previously had evidence of active tuberculosis and did not receive appropriate and documented treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- China (3):
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Second Affiliate Hospital of Zhejiang Medical University, Hangzhou, Zhejiang
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University, Shanghai

REFERENCES:
- [Derived] Zheng M, Chen X, Wang F, Chen J, Jackson K, Yang F, Payne C, Li H, Wang Y, Xiao Z, Zheng J. Pharmacokinetics, Safety, and Efficacy of Ixekizumab in Chinese Patients with Moderate-to-Severe Plaque Psoriasis: A Phase 1, Single- and Multiple-Dose Study. Adv Ther. 2023 Sep;40(9):3804-3816. doi: 10.1007/s12325-023-02575-1. Epub 2023 Jun 25. PMID 37356077

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All the re-enrolled participants from single dose period (SDP) to multiple dose period (MDP) have been washed out and screened for eligibility to MDP.
Groups:
- Ixekizumab 80mg Q2W Multiple Dose: Participants received multiple doses of Ixekizumab starting with 160mg initial dose followed by 80mg every two weeks (Q2W) by subcutaneous injection.
- Ixekizumab 80mg Q4W Multiple Dose: Participants received multiple doses of 80mg Ixekizumab starting with 160mg initial dose followed by 80mg every four weeks (Q4W) by subcutaneous injection.
Period: Single Dose Period
Arm/Group | Ixekizumab Single Dose | Ixekizumab 80mg Q2W Multiple Dose | Ixekizumab 80mg Q4W Multiple Dose
Started | 12 | 0 | 0
Completed | 12 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Multiple Dose Period
Arm/Group | Ixekizumab Single Dose | Ixekizumab 80mg Q2W Multiple Dose | Ixekizumab 80mg Q4W Multiple Dose
Started | 0 | 14 (Participants who completed single dose had option to enroll into multiple dose.) | 15 (Participants who completed single dose had option to enroll into multiple dose.)
Participants Enrolled From Single Dose | 0 | 7 | 2
Completed | 0 | 14 | 14
Not Completed | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All the re-enrolled participants from SDP to MDP have been washed out and screened for eligibility to MDP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixekizumab Single Dose | Ixekizumab 80mg Q2W Multiple Dose | Ixekizumab 80mg Q4W Multiple Dose | Total
Number analyzed (Participants) | 12 | 14 | 15 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: All the re-enrolled participants from SDP to MDP have been washed out and screened for eligibility to MDP.
  years
    Single Dose: number analyzed (Participants) | 12 | 0 | 0 | 12
    Single Dose | 49.0 (12.1) |  |  | 49.0 (12.1)
    Multiple Dose: number analyzed (Participants) | 0 | 14 | 15 | 29
    Multiple Dose |  | 45.6 (12.5) | 45.5 (16.1) | 45.6 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All the re-enrolled participants from SDP to MDP have been washed out and screened for eligibility to MDP.
  Participants
    Single Dose: number analyzed (Participants) | 12 | 0 | 0 | 12
    Single Dose: Female | 2 | 0 | 0 | 2
    Single Dose: Male | 10 | 0 | 0 | 10
    Multiple Dose: number analyzed (Participants) | 0 | 14 | 15 | 29
    Multiple Dose: Female | 0 | 3 | 5 | 8
    Multiple Dose: Male | 0 | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All the re-enrolled participants from SDP to MDP have been washed out and screened for eligibility to MDP.
  Participants
    Single Dose Phase: number analyzed (Participants) | 12 | 0 | 0 | 12
    Single Dose Phase: Hispanic or Latino | 0 | 0 | 0 | 0
    Single Dose Phase: Not Hispanic or Latino | 12 | 0 | 0 | 12
    Single Dose Phase: Unknown or Not Reported | 0 | 0 | 0 | 0
    Multiple Dose Phase: number analyzed (Participants) | 0 | 14 | 15 | 29
    Multiple Dose Phase: Hispanic or Latino | 0 | 0 | 0 | 0
    Multiple Dose Phase: Not Hispanic or Latino | 0 | 14 | 15 | 29
    Multiple Dose Phase: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All the re-enrolled participants from SDP to MDP have been washed out and screened for eligibility to MDP.
  Participants
    Single Dose Phase: number analyzed (Participants) | 12 | 0 | 0 | 12
    Single Dose Phase: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Single Dose Phase: Asian | 12 | 0 | 0 | 12
    Single Dose Phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Single Dose Phase: Black or African American | 0 | 0 | 0 | 0
    Single Dose Phase: White | 0 | 0 | 0 | 0
    Single Dose Phase: More than one race | 0 | 0 | 0 | 0
    Single Dose Phase: Unknown or Not Reported | 0 | 0 | 0 | 0
    Multiple Dose Phase: number analyzed (Participants) | 0 | 14 | 15 | 29
    Multiple Dose Phase: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Multiple Dose Phase: Asian | 0 | 14 | 15 | 29
    Multiple Dose Phase: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Multiple Dose Phase: Black or African American | 0 | 0 | 0 | 0
    Multiple Dose Phase: White | 0 | 0 | 0 | 0
    Multiple Dose Phase: More than one race | 0 | 0 | 0 | 0
    Multiple Dose Phase: Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China: Single Dose | 12 | 0 | 0 | 12
  China: Multiple Dose | 0 | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Ixekizumab (Single Dose)
Description: Pharmacokinetics (PK): Cmax is the maximum observed concentration of Ixekizumab into serum.
Time Frame: Single dose: Predose, day 1, 3, 5, 8, 11, 15, 22, 29, 43, 57, 85, 113, 141
Population: All randomized participants who received at least one dose of Ixekizumab in single dose group and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Arm/Group | Ixekizumab Single Dose
Number analyzed (Participants) | 12
Microgram per milliliter (ug/mL) | 6.90 (43)

2. Primary Outcome: Pharmacokinetics: Area Under Concentration From Time Zero to Infinity (AUC 0toinf) of Ixekizumab (Single Dose)
Description: Pharmacokinetics: Area Under the Concentration Versus Time Curve (AUC) from time zero to infinity was reported.
Time Frame: Predose, day 1, 3, 5, 8, 11, 15, 22, 29, 43, 57, 85, 113, 141
Population: All randomized participants who received at least one dose of Ixekizumab in single dose group and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*day per milliliter (ug*day/mL)
Arm/Group | Ixekizumab Single Dose
Number analyzed (Participants) | 12
Microgram*day per milliliter (ug*day/mL) | 147 (48)

3. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Ixekizumab (Multiple Dose)
Description: Pharmacokinetics: Cmax is the maximum observed concentration of Ixekizumab into serum.
Time Frame: day 57 (pre-dose), 59, 61, 64, 67, 71, 78, 85, 99, 113, 141, 169, 197
Population: All randomized participants who received at least one dose of Ixekizumab in multiple dose group and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Arm/Group | Ixekizumab 80mg Q2W Multiple Dose | Ixekizumab 80mg Q4W Multiple Dose
Number analyzed (Participants) | 14 | 14
Microgram per milliliter (ug/mL) | 19.9 (27) | 13.4 (32)

4. Primary Outcome: Pharmacokinetics: Area Under Concentration From Time Zero to 336h (AUC 0 to 336h) of Ixekizumab (Multiple Dose)
Description: Pharmacokinetics: Area under concentration of Ixekizumab from time Zero to 336h (AUC 0 to 336h) was reported (Multiple dose).
Time Frame: day 57 (Pre-dose), 59, 61, 64, 67, 71
Population: All randomized participants multiple dose period who received at least one dose of Ixekizumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*day per milliliter (ug*day/mL)
Arm/Group | Ixekizumab 80mg Q2W Multiple Dose | Ixekizumab 80mg Q4W Multiple Dose
Number analyzed (Participants) | 14 | 14
Microgram*day per milliliter (ug*day/mL) | 224 (25) | 136 (31)

5. Primary Outcome: Pharmacokinetics: Area Under Concentration From Time Zero to 672h (AUC 0 to 672h) of Ixekizumab (Multiple Dose)
Description: Pharmacokinetics: Area under concentration of Ixekizumab from time zero to 672h (AUC 0 to 672h) was reported (Multiple dose).
Time Frame: day 57 (Pre-dose), 59, 61, 64, 67, 71, 78, 85
Population: All randomized participants in Ixekizumab Q4W arm who received at least one dose of Ixekizumab and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*day per milliliter (ug*day/mL)
Arm/Group | Ixekizumab 80mg Q4W Multiple Dose
Number analyzed (Participants) | 14
Microgram*day per milliliter (ug*day/mL) | 213 (29)

ADVERSE EVENTS:
Time Frame: Baseline to end of the study (up to 20 weeks)
Description: All Randomized participants.
Arm/Group | Ixekizumab Single Dose | Ixekizumab 80mg Q2W Multiple Dose | Ixekizumab 80mg Q4W Multiple Dose
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/14 | 0/15
Other Adverse Events (participants affected / at risk) | 11/12 | 11/14 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab Single Dose (N=12) | Ixekizumab 80mg Q2W Multiple Dose (N=14) | Ixekizumab 80mg Q4W Multiple Dose (N=15)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixekizumab Single Dose (N=12) | Ixekizumab 80mg Q2W Multiple Dose (N=14) | Ixekizumab 80mg Q4W Multiple Dose (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Dental discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (5) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (2) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (2) | 1 (1)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea manuum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Echocardiogram abnormal (Investigations) | 0 (0) | 1 (1) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1) | 3 (4) | 2 (2)
Glucose urine present (Investigations) | 0 (0) | 1 (3) | 0 (0)
Low density lipoprotein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Protein urine present (Investigations) | 4 (4) | 2 (4) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 1 (1) | 1 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 2 (4)
White blood cells urine positive (Investigations) | 0 (0) | 1 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (4) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (5) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Menstruation delayed (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nail psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (10) | 2 (3)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-06-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03073213/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT03073213/SAP_001.pdf